CLINICAL TRIAL: NCT03937310
Title: What is the Role of Next-generation Sequencing in Non-union of Orthopaedic Cases
Brief Title: NGS for Non-unions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: Krieg2019
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Nonunion of Fracture
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical intervention for non-union: The investigation group will consist of cases undergoing surgical intervention for non-union
  Interventions: Diagnostic Test: Next-generation sequencing of swabs collected during surgery
- Acute fracture fixation: The control group will consist of cases undergoing acute fracture fixation
  Interventions: Diagnostic Test: Next-generation sequencing of swabs collected during surgery

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing of swabs collected during surgery — Traditional swabs for culturing as well as swabs for NGS testing will be collected

SUMMARY:
The purpose of this study is to investigate the role of genetic testing to look for possible infection as a cause for failure of non-healing fractures. The study aims to compare the results of genetic testing known as NGS to standardized clinical laboratory tests for diagnosing infections to see if NGS may be a better diagnostic tool.

ELIGIBILITY:
Investigational group:

Inclusion:

1. Patients undergoing open biopsy / surgical intervention for nonunion following a traumatic (open or closed) long bone fracture (femur shaft, tibia, humerus) which was initially treated operatively.Inclusion Criteria:
2. Nonunions will be defined as a failure to progress towards expected union within an anticipated timeframe, and this judgment will be made by the attending caring for each patient. No specific timeframe or arbitrary cut points will be defined to allow for the considerable variation in fracture healing and different anatomical sites.
3. Presumed Septic and Aseptic nonunions
4. >18 years old and able to provide informed consent

Exclusion Criteria:

Exclusion:

1. Pathological fractures at index injury
2. Patients on antibiotic therapy <2 weeks prior to surgery

INCLUSION/ EXCLUSION CRITERIA FOR CONTROL GROUP:

Inclusion:

1. Patients undergoing surgical intervention for nonunion following a traumatic closed long bone fractures (femur shaft, tibia, humerus)
2. >18 years old and able to provide informed consent

Exclusion:

1. Pathological fractures at index injury
2. Patients on antibiotic therapy <2 weeks prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be chosen based on intervention planned. This is not an interventional study, just an observational study
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-01-03 (Estimated); Study Completion 2022-02-03 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 6 months post-op
  Need for additional re-operation or intervention within follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States